CLINICAL TRIAL: NCT02525107
Title: Omega 3 Fatty Acid Therapy for Prevention of Vaso-occlusive Crisis and Manifestations in Omani Patients With Sickle Cell Disease
Brief Title: Prevention of Vaso-occlusive Painful Crisis by Using Omega-3 Fatty Acid Supplements
Acronym: OM3FA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sultan Qaboos University (Other)
Collaborators: Ministry of Health, Sultanate of Oman (Unknown); London Metropolitian University (Unknown)
Responsible Party: Principal Investigator, Salam Alkindi, Professor & Head, Department of Haematology, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORG/HSS/14/013
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Sickle Cell Disease
Keywords: Prevention of Vaso Occlusive Painful Crisis
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCD patients on Hydroxyurea (Experimental): Omega-3 capsules [750 mg], 4 capsules a day for 52 weeks. [Each capsule will contain 417.9mg Docosahexaenoic acid [DHA], 50.8 mg Eicosapentaenoic acid [EPA] and 11.9mg Arachidonic acid [AA] and 1000 IU Vitamin E]
  Interventions: Dietary Supplement: Omega-3 capsules; Dietary Supplement: Placebo
- SCD patients not on Hydroxyurea (Experimental): Dietary Supplement: Placebo [730 mg], 4 capsules a day for 52 weeks.[Each capsule will contain 538.2mg Oleic Acid [OA] and 1000 IU Vitamin E]
  Interventions: Dietary Supplement: Omega-3 capsules; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 capsules — SCD patients on Hydroxyurea
  Other Names: Omega-3 Fatty acid, fish oil supplement
  Arms: SCD patients on Hydroxyurea
Dietary Supplement: Placebo — SCD patients on Hydroxyurea
  Arms: SCD patients on Hydroxyurea
Dietary Supplement: Omega-3 capsules — SCD patients not on Hydroxyurea
  Other Names: Omega-3 Fatty acid, fish oil supplement
  Arms: SCD patients not on Hydroxyurea
Dietary Supplement: Placebo — SCD patients not on Hydroxyurea
  Arms: SCD patients not on Hydroxyurea

SUMMARY:
140 SCD patients [70 on Hydroxyurea] will receive Omega-3 capsules whereas another 140 SCD patients [70 on Hydroxyurea] will receive placebo and will be recruited from the Sultan Qaboos University Hospital [SQUH] haematology specialty clinics. Patients will be randomized in a 1:1 ratio to receive placebo or Omega-3 for 52 weeks. The aim is to investigate the therapeutic potential of omega-3 fatty acids in the prevention of vaso-occlusive crisis in Omani patients with sickle cell disease[SCD].

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Sickle cell disease patients.
* Patients already receiving Hydroxyurea[HU] are eligible for the study.
* Patients able and willing to comply with the procedures in the study protocol.

Exclusion Criteria:

* Acute episodes (infection, vaso-occlusive crises (VOC), acute chest syndrome (ACS), stroke, priapism, splenic sequestration) in the past one month before enrolment.
* Previous stroke, and other co-morbid diseases like Essential Hypertension, Cardiomyopathy and Heart failure, Diabetes, Chronic Renal Failure.
* Patients with a history of adverse reaction to omega-3 fatty acid supplementation.
* Blood transfusion in the previous 3 months.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of VOC | 52 weeks
  Reduction of the number of Emergency and Hospital visits for VOC episodes compared to the previous 52 weeks
Severity of VOC | 52 weeks
  Reduction in the average visual analog score for pain with scores ranging from 0[no pain] to 10[worst possible pain] recorded during VOC episodes compared to the previous 52 weeks
Duration of Hospitalization | 52 weeks
  Reduction in the number of days in hospital with VOC pain compared to the previous 52 weeks

SECONDARY OUTCOMES:
Red blood cells membrane fatty acids profile | 52 weeks
  Measurement of red blood cell membrane ethanolamine phosphoglyceride[DHA, EPA, AA] at baseline and after 52 weeks intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, Sultan Qaboos University, Muscat, Oman